CLINICAL TRIAL: NCT03793205
Title: Long-acting Granulocyte Colony Stimulating Factor for the Prevention of Febrile Neutropenia in Gynecologic Cancer Patients: A Prospective Cohort Study
Brief Title: G-CSF for the Prevention of Febrile Neutropenia in Gynecologic Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GO-GCSF
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Gynecologic Cancer; Myelosuppression Adult; Febrile Neutropenia; Chemotherapy-induced Neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Intervention Model Description: After the chemotherapy, patients accepted long-acting G-CSF and/or short-acting G-CSF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-acting G-CSF group (Experimental): Patients in long-acting G-CSF group accept long-acting with or without short-acting G-CSF.
  Interventions: Drug: Long-acting G-CSF
- Short-acting G-CSF group (Experimental): Patients in long-acting G-CSF group only accept short-acting G-CSF.
  Interventions: Drug: Short-acting G-CSF

INTERVENTIONS:
Drug: Long-acting G-CSF — Long-acting G-CSF will be given 48 hours after the chemotherapy. A supplement of short-acting G-CSF will be given as required.
  Arms: Long-acting G-CSF group
Drug: Short-acting G-CSF — Short-acting G-CSF will be given as required 24 hours after the chemotherapy.
  Arms: Short-acting G-CSF group

SUMMARY:
This study aims to analyze the effects of long-acting granulocyte colony stimulating factor (G-CSF) on the prevention febrile neutropenia (FN) in gynecologic cancer patients. Patients all accepted platinum-based chemotherapy 3-4 weeks once per course. The primary end is the incidence of FN in every course of chemotherapy. After the chemotherapy, patients accepted long-acting G-CSF and/or short-acting G-CSF. The secondary ends include: the incidences of myelosuppression, doses of G-CSF and its expenses, visits to outpatient and emergency clinics, adverse events related to G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary gynecologic cancer
* Good performance status
* Aged 18 years or older
* Signed an approved informed consents
* No immunosuppressive disease

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia | One year
  Incidence of febrile neutropenia in each course

SECONDARY OUTCOMES:
Incidences of grade 3/4 myelosuppression | One year
  Incidences of grade 3/4 myelosuppression in each course
Times of visits to outpatient and emergency clinics | One year
  Visits to outpatient and emergency clinics in each course
Doses of G-CSF | One year
  Doses of G-CSF administrated in each course

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen X, Wu M, Ma S, Tan X, Zhong S, Li L. Effects of long-acting versus short-acting granulocyte colony stimulating factor after radiotherapy in gynecologic malignancies: a prospective observational cohort study. BMC Cancer. 2024 Dec 18;24(1):1512. doi: 10.1186/s12885-024-13296-1. PMID 39696092